CLINICAL TRIAL: NCT00934804
Title: Accuracy of the Galilei Analyzer to Calculate the Effective Corneal Power After Corneal Refractive Surgery
Acronym: Galilei
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator separating employment from University.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19183
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2009-10

CONDITIONS: Cataracts
Keywords: refractive surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparative Diagnostic system (Experimental): Galilei dual Scheimpflug analyzer
  Interventions: Device: Galilei dual Scheimpflug analyzer

INTERVENTIONS:
Device: Galilei dual Scheimpflug analyzer — The Galilei dual Scheimpflug analyzer is a non-invasive, diagnostic system that combines dual rotating Scheimpflug camera measurements and Placido optical system for corneal topography and 3D analysis of the anterior eye segment.
  Other Names: Holladay I, HofferQ, SRKT

SUMMARY:
The purpose of this study is to determine the accuracy of the Galilei corneal analyzer to calculate the effective corneal power (keratometry, corneal curvature) in patients who have undergone both corneal refractive surgery and lens extraction with intraocular lens implantation.

DETAILED DESCRIPTION:
The accuracy of IOL calculation is important for the visual outcome of patients undergoing cataract extraction and IOL implantation. Different formulas such as Holladay I, HofferQ, SRKT have been used with excellent results. All formulas use the corneal power among other factors to calculate the IOL power. Corneal refractive surgery i.e. radial keratotomy (RK), photorefractive keratectomy (PRK), and Laser in situ keratomileusis (LASIK) changes the corneal power; therefore, it is difficult to measure the true corneal power after surgery by any form of direct measurement, such as keratometry, or corneal topography. Keratometry and topography assume a normal relationship between the anterior and posterior corneal curvatures, and measure the anterior corneal radius. RK for myopia flattens both the anterior corneal radius and the posterior corneal radius while PRK and LASIK for myopia flattens the anterior corneal radius but leaves the posterior corneal radius mostly unchanged.

Standard keratometry measures an intermediate area and extrapolates the central power based on some very broad assumptions. For this reason, keratometry, autokeratometry and simulated keratometry by topography will typically over-estimate central corneal power following keratorefractive surgery for myopia. This inaccuracy leads to an inability to meet the patients' rising expectations and with the increasing popularity of refractive surgery, calculating intraocular lens (IOL) power after refractive surgery is becoming increasingly important.

Different methods to calculate the effective corneal power (keratometry) after refractive surgery have been described (historical data, effective refractive power, modified Maloney method, etc), however, intraocular lens power calculations in eyes with previous refractive surgery remains difficult because of the inaccuracy of keratometry power measurements.

The Galilei dual Scheimpflug analyzer is a non-invasive, diagnostic system that combines dual rotating Scheimpflug camera measurements and Placido optical system for corneal topography and 3D analysis of the anterior eye segment. It provides pachymetry as well as elevation and curvature mapping of the cornea. Additionally, the Ray tracing system delivers a more accurate total corneal power and anterior chamber depth. The total corneal power that the Galilei provides is an alternative that seems to be more accurate to calculate the IOL power in patients who have undergone keratorefractive surgery prior to cataract extraction and IOL implantation.

The purpose of this study is to determine the accuracy of the Galilei to calculate the effective corneal power (keratometry, corneal curvature) in patients who have undergone both corneal refractive surgery and lens extraction with intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects MUST fulfill the following conditions to qualify for enrollment into the trial:

  * Subject must have undergone corneal refractive surgery (RK, PRK or LASIK) prior to cataract extraction.
  * Age: 40 to 80 years old.
  * Subjects must have undergone cataract extraction at least 4 weeks prior to enrollment in this trial.
  * Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

Subjects with ANY of the following conditions on the eligibility exam may NOT be enrolled into the trial.

Preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphtalmus or macrophtalmus, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.

Uncontrolled diabetes. Use of any systemic or topical drug known to interfere with visual performance. Contact lens use during the active treatment portion of the trial. Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.

Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.

Intraocular conventional surgery (other than cataract extraction) within the past three months or intraocular laser surgery within one month in the operated eye.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Galilei to calculate the effective corneal power (keratometry, corneal curvature) in patients who have undergone both corneal refractive surgery and lens extraction with intraocular lens implantation. | Three Months

CONTACTS AND LOCATIONS:
Overall Officials: Helga P. Sandoval, MD, Principal Investigator — Medical University of South Carolina, Storm Eye Institute
Locations (1):
- Helga Sandoval, MD, Charleston, South Carolina, United States